CLINICAL TRIAL: NCT06759233
Title: Endoscopic Cryoablation Combined With PD-1 in Advanced Gastric Cancer and Its Immune Activation Mechanism Study
Brief Title: Endoscopic Cryoablation Combined With PD-1 in Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhongguang Luo, MD (Other)
Responsible Party: Sponsor-Investigator, Zhongguang Luo, MD, Chief Physician, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-1042
Record Dates: First submitted 2024-09-19; First posted 2025-01-06 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer
Keywords: ECAT; PD-1
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- endoscopic cryoballoon ablation treatment（ECAT）+ PD-1 (Experimental): Patients with advanced gastric cancer enrolled in the study will undergo ECAT (endoscopic cryoballoon ablation treatment). Within three days before or after ECAT treatment, they will receive the first dose of PD-1 monoclonal antibody therapy as part of this study (the dosing schedule for PD-1 therapy will follow the drug's prescribing information).
  Interventions: Procedure: endoscopic cryoballoon ablation treatment(ECAT)+PD-1

INTERVENTIONS:
Procedure: endoscopic cryoballoon ablation treatment(ECAT)+PD-1 — ECAT: A cryoballoon with catheter is inserted along the endoscopic forceps channel, the balloon is placed on the surface of the tumor, and the balloon is dilated so that it fits snugly over the lesion. The freezing cycle is initiated and continued for 2-3 minutes, and then the balloon is rewarmed and frozen again for 2-3 minutes; the freeze-rewarm cycle is repeated twice.
  PD-1:The first PD-1 monoclonal antibody treatment in this study was given within 3 days before and after ECAT treatment, and subsequent treatment was given every three weeks according to the instructions.

SUMMARY:
To clarify the efficacy and safety of endoscopic cryoablation combined with PD-1 monoclonal antibody treatment regimen in advanced gastric cancer.

DETAILED DESCRIPTION:
This study is a single-center, single-arm, self-controlled, experimental, non-randomized exploratory clinical trial, aiming to enroll 15 patients with advanced gastric cancer. Each enrolled patient will be assigned a case number. This case number, along with the patient's name initials, will be recorded on every page of the case report form (CRF). Enrolled patients will receive local gastric ECAT (endoscopic cryoballoon ablation treatment) combined with PD-1 monoclonal antibody therapy for the evaluation of efficacy and safety, as well as immunological assessments of peripheral circulation and local tumor tissue. Patients will be followed during the treatment period and for six months after treatment termination for study observation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with advanced gastric cancer (stage IV in AJCC 8th edition staging, including locally progressive gastric cancer with unresectable factors (IVa) and gastric cancer with distant metastases (IVb); Bowman's staging type I, II, and III), who are unable to be surgically resected or do not tolerate surgical resection, and who have undergone progression after 1-2 lines of conventional chemotherapy;
2. Age greater than 18 years and less than 80 years;
3. WHO pathology type: adenocarcinoma, neuroendocrine tumor;
4. Expected survival greater than 3 months and controllable distant metastases as judged by the physician;
5. Important organ functions must be met: ① Liver function: ALT and AST ≤ 2.5 times the positive range, total bilirubin ≤ 2.0mg/dL; ② Renal function: creatinine clearance ≥ 40mL/min calculated using the EPI formula;
6. Blood routine: Hgb≥70g/L,ANC≥1.5×109/L,PLT≥80×109/L;
7. Coagulation function: PT and APPT <2 times the normal value;
8. Pregnancy test must be negative in women of childbearing age;
9. ECOG score ≤2;
10. Signed informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women with pregnancy plans within six months;
2. Infectious diseases (e.g. AIDS, syphilis, active tuberculosis);
3. Patients with active hepatitis B or C infection;
4. Combination of other primary malignant tumors;
5. Patients who have participated in a clinical trial within one month;
6. Patients taking antiplatelet or anticoagulant drugs within the last week;
7. Patients with gastric cancer combined with active bleeding;
8. Large amount of ascites (ascites ≥3000ml);
9. Cardia obstruction or pyloric obstruction;
10. patients with combined active infection or autoimmune disease;
11. Those who the doctor thinks there are other reasons not to be included in the treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to study completion, assessed up to 2 years
  PFS is measured from the start of treatment until the first documented evidence of disease progression (based on RECIST 1.1) or death from any cause, whichever occurs first.
Overall-Survival (OS) | From enrollment to study completion, assessed up to 5 years
  The length of time from the start of treatment until death from any cause.

SECONDARY OUTCOMES:
Percentage of participants achieving complete remission (CR) and partial remission (PR) after treatment | 3 to 24 weeks after the end of treatment
  Objective remission rate (ORR), the percentage of participants whose tumors shrink by a certain amount and remain there for a certain period of time, including complete remission (CR) and partial remission (PR). CR (Complete remission): Complete disappearance of the target lesion, with no new lesions produced, and lasting for more than 4 weeks. PR (Partial remission): the sum of the largest diameters of the target lesions is reduced by more than 30%, and lasts for more than 4 weeks.
Percentage of participants achieving remission (PR+CR) and lesion stabilization (SD) after treatment | 3 to 24 weeks after the end of treatment
  Disease control rate (DCR) is the percentage of participants who achieve remission (PR+CR) and stabilization of lesions (SD) after the treatment. Stable disease (SD) means that the sum of the largest diameters of the tumor lesions has not shrunk to PR, or has not enlarged to PD.
Number of participants with treatment-related adverse events | From the start of treatment to 24 weeks after the end of treatment
  The number of patients who experience ECAT-related adverse events (such as intraoperative bleeding, intraoperative perforation, postoperative bleeding, etc.)

OTHER OUTCOMES:
Number of immune cells in peripheral blood | From enrollment to study completion, assessed up to 24 weeks
  Peripheral blood will be analyzed for the number of immune cells after applying flow cytometry and mRNA sequencing.
Number of immune cells in tumor tissues | From enrollment to study completion, assessed up to 24 weeks
  Apply mRNA sequencing, immunohistochemistry and immunofluorescence to analyze the number of immune cells in tumor tissues, including CTL, Treg, DC, TAM, MDSC, NK, NKT and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, China